CLINICAL TRIAL: NCT03227458
Title: DHEA Augmentation of Musculoskeletal Adaptations to Exercise in Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16-2427; 5R01AG053489-05 (NIH)
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Low Bone Mass; Osteoporosis, Postmenopausal
Keywords: areal bone mineral density; dehydroepiandrosterone (DHEA); postmenopause; exercise; sex hormones
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Motor Activity | interventions — Dehydroepiandrosterone; Exercise

STUDY DESIGN:
Intervention Model Description: All participants will take 1 study pill (50 mg DHEA or placebo: double-blinded) daily for 36 weeks. The research pharmacist will dispense study drug according to the randomization code and maintain drug dispensation records, which will be monitored by the study biostatistician. Two-thirds of participants will engage in bone-loading exercise 3 days per week for the 36 weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study drug will be masked. 50 mg DHEA or placebo: double-blinded. Exercise will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise and DHEA (Active Comparator): 1 study pill containing 50 mg of DHEA daily for 36 weeks and supervised bone-loading exercise on 3 days per week for 36 weeks.
  Interventions: Other: DHEA; Behavioral: Exercise
- Exercise and Placebo (Active Comparator): 1 study pill containing placebo daily for 36 weeks and supervised bone-loading exercise on 3 days per week for 36 weeks.
  Interventions: Other: Placebo; Behavioral: Exercise
- DHEA only (Active Comparator): 1 study pill containing 50 mg of DHEA daily for 36 weeks
  Interventions: Other: DHEA

INTERVENTIONS:
Other: DHEA — Participants will take 1 study pill (50 mg DHEA) daily for 36 weeks.
  Other Names: DHEA therapy
  Arms: DHEA only; Exercise and DHEA
Other: Placebo — Participants will take placebo daily for 36 weeks.
  Arms: Exercise and Placebo
Behavioral: Exercise — bone-loading exercise on 3 days per week for 38 weeks
  Other Names: bone-loading exercise
  Arms: Exercise and DHEA; Exercise and Placebo

SUMMARY:
To determine whether the musculoskeletal adaptations to bone-loading exercise can be significantly augmented in older women (aged 60-85) with low bone mass (osteopenia; T-scores <-1.0 and >-2.5) or moderate osteoporosis (T-scores < -2.5 and >= -3.0) and by restoring serum DHEAS to young adult levels by oral DHEA replacement.

DETAILED DESCRIPTION:
This will be the first study to measure changes in areal bone mineral density (aBMD) and fat-free mass (FFM) in response to dehydroepiandrosterone (DHEA) alone and combined with exercise in postmenopausal women. The body of evidence from carefully executed Randomized Controlled Studies (RCTs) provides support for DHEA therapy to increase aBMD and FFM in older women. Less is known about whether DHEA therapy enhances the effects of exercise on the aging musculoskeletal system when an appropriate mechanical stimulus is applied.

ELIGIBILITY:
Inclusion Criteria:

* non-frail, as determined by short physical performance battery (SPPB) score > 9 (0-12 scale);
* 5 years or longer since menopause (defined as last menstrual period);
* willing to participate in a 36-week exercise program that will start at a moderate intensity and gradually progress to a higher intensity;
* willing to be randomized to an exercise or a no-exercise arm of the study;
* willing to take DHEA (50mg/d) or a placebo pill daily and remain blinded for up to 36 weeks;
* not performing resistance exercise training or high impact weight-bearing exercise (e.g., jogging) ≥ 2 days per week in the past 6 months;
* ambulatory without assistive devices;
* serum DHEAS < 140 μg/dL (3.8 μmol/L);
* low bone mass or moderate osteoporosis defined as lumbar spine or proximal hip aBMD t-scores < -1.0 and > = -3.0;
* refusal of standard osteoporosis treatment in women with moderate osteoporosis (BMD t-scores >=-3.0 and =< 2.5).
* evidence of a negative (no findings suspicious for breast cancer) mammogram within the past 12 months;
* planning to reside in the Denver area for the duration of the study
* normal cognitive function, as determined by a Mini-Cog score > = 4

Exclusion Criteria:

* history of hospitalization for Corona Virus Disease-19 (COVID-19)
* does not meet Centers for Disease Control and Prevention (CDC) recommendations for home isolation because has had a positive severe acute respiratory syndrome corona virus-2 (SARS-COV-2) test less than 10 days before study entry; or has had fever within the past 3 days and respiratory symptoms have not improved; or symptoms first appeared less than 10 days before study entry
* uncontrolled hypertension defined as resting systolic blood pressure (sBP) >150 mmHg or diastolic blood pressure (dBP) >90 mmHg; participants who do not meet these criteria at first screening will be re-evaluated, including follow-up evaluation by their Primary Care Physician (PCP) with initiation or adjustment of anti-hypertensive medications;
* diagnosed ischemic heart disease or indicators of unstable ischemic heart disease (e.g., angina, ST segment depression) or arrhythmias at rest or during the Gated Exercise Test (GXT) without negative follow-up evaluation will be cause for exclusion; follow-up evaluation must include diagnostic testing (e.g., thallium stress test) with interpretation by a cardiologist;
* diagnosis of heart failure, clinically significant aortic stenosis, uncontrolled angina, or uncontrolled arrhythmia.
* pulmonary disease requiring use of oral steroids within the previous 6 months or the use of supplemental oxygen ≥ 4 liters with physical exertion
* orthopedic problems (e.g., severe osteoarthritis, rheumatoid arthritis) that greatly limit the ability to perform moderate to high intensity resistance exercise (e.g., unable to be properly positioned in exercise equipment or to have severely restricted range of motion even after modifications have been made)
* hip fracture, hip or knee replacement, or spinal surgery in the past 6 months;
* undergoing physical therapy involving the lower extremities;
* hematocrit (HCT) > 54%;
* thyroid dysfunction, defined as an ultrasensitive thyroid stimulating hormone (TSH) < 0.4 or > 10.0 microunits/mL;, without signs or symptoms of clinical hypo- or hyperthyroidism. Volunteers with abnormal TSH values will be re-considered for participation in the study after follow-up evaluation by their PCP with initiation or adjustment of thyroid hormone replacement;
* acute liver disease indicated by liver function tests (alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase) ≥ 1.5 times the upper limits of normal;
* estimated glomerular filtration rate (eGFR) < 45, using the Modification of Diet in Renal Disease (MDRD) equation (Levey et al, Annals Inter Med, 1999; Munter et al, Clin J Am Soc Nephrology, 2009);
* poorly controlled diabetes mellitus based on HbA1c > 8.5%, or use of insulin;
* fasted serum triglycerides > 400 mg/dL;
* serum 25-hydroxy vitamin D <20 ng/mL; volunteers will be re-considered for participation in the study after follow-up evaluation by their PCP with initiation or adjustment of vitamin D supplementation per the study's vitamin D repletion protocol.
* use of DHEA supplementation or sex hormones in the past 6 months. Use of prescription low dose vaginal estrogen creams (Premarin or Estrace) 3 days per week will not be exclusionary.
* use in the past 6 months of any medications known to alter bone metabolism (e.g., oral glucocorticoids, bone anti-resorptive agents);
* documented history of cognitive impairment or dementia, or Mini-Cog < 4;
* current smoker;
* personal history of breast, ovarian, metastatic endometrial, or cervical cancer;
* any cancer requiring treatment in the past 3 years except non-melanoma skin cancers;
* un-diagnosed vaginal bleeding;
* women who, in the judgment of the study physician, appear incapable of safely participating in the exercise (e.g., neuromuscular/musculoskeletal impairment)
* use of insulin;
* lumbar spine, total hip, or femoral neck aBMD t-scores < -3.0;
* secondary osteoporosis

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Change in lumbar spine aBMD | Baseline and 36 Weeks
  mean change from baseline in lumbar spine aBMD

SECONDARY OUTCOMES:
Change in total hip aBMD | 36 Weeks
  mean change from baseline in total hip aBMD
Change in regional hip aBMD | Baseline and 36 Weeks
  mean change from baseline in regional hip aBMD
Change in Vertebral (L1-2) total volumetric bone mineral density (vBMD) | Baseline and 36 Weeks
  mean change from baseline in vertebral total volumetric BMD
Change in Vertebral (L1-2) cortical vBMD | Baseline and 36 Weeks
  mean change from baseline in vertebral cortical volumetric BMD
Change in Vertebral (L1-2) trabecular vBMD | Baseline and 36 Weeks
  mean change from baseline in vertebral trabecular volumetric BMD
Change in Femoral total vBMD | Baseline and 36 Weeks
  mean change from baseline in femoral total volumetric BMD
Change in Femoral cortical vBMD | Baseline and 36 Weeks
  mean change from baseline in femoral cortical volumetric BMD
Change in Femoral trabecular vBMD | Baseline and 36 Weeks
  mean change from baseline in femoral trabecular volumetric BMD
Change in Vertebral (L1-2) strength, stance model | Baseline and 36 Weeks
  mean change from baseline in the estimated strength of L1-2 vertebrae in a stance model
Change in Vertebral (L1-2) strength, fall model | Baseline and 36 Weeks
  mean change from baseline in the estimated strength of L1-2 vertebrae in a fall model
Change in Proximal femur strength, stance model | Baseline and 36 Weeks
  mean change from baseline in the estimated strength of the proximal femur in a stance model
Change in Proximal femur strength, fall model | Baseline and 36 Weeks
  mean change from baseline in the estimated strength of the proximal femur in a fall model
Change in Total body fat-free mass | Baseline and 36 Weeks
  mean change from baseline in total body fat-free mass

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Jankowski, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No